CLINICAL TRIAL: NCT05872334
Title: Exploratory Clinical Trial for Evaluating the Safety and Efficacy of MONOFIX® on Fascial Closure of Mid-line Wound for Patients With Colon Cancer Underwent Minimally Invasive Surgery: Single-center, Non-blinded, and Single-arm Design
Brief Title: The Safety and Feasibility of MONOFIX on Fascial Closure of Mid-line Wound After Minimally Invasive Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Woo Yong Lee, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MONOFIX_01
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Colon Cancer; Rectal Cancer; Colon Adenocarcinoma; Rectal Adenocarcinoma
Keywords: minimally invasive surgery; Barbed suture
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monofix (Experimental): In patients who underwent laparoscopic colorectal cancer surgery, the fascial closure of the midline incision was performed using a running suture type with Monofix, one of the barbed sutures.
  Interventions: Device: Monofix
- Control group (No Intervention): In patients who underwent laparoscopic colorectal cancer surgery, the fascial closure of the midline incision was performed using an interrupted suture type with PDS-II, one of the monofilament sutures.

INTERVENTIONS:
Device: Monofix — a new absorbable barbed suture device
  Arms: Monofix

SUMMARY:
This clinical trial aims to evaluate the safety and feasibility of mid-line fascial suturing using MONOFIX sutures in patients undergoing minimally invasive surgery for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenocarcinoma
* Elective (or planned) curative surgery
* Laparoscopic surgery
* Midline incision less than 10 cm

Exclusion Criteria:

* Previous laparotomy with midline incision more than 10cm.
* Systemic chemotherapy for any cause within the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Incisional hernia | 18 months from surgery
  Incisional hernia diagnosed by CT scan.

SECONDARY OUTCOMES:
Wound infection | 1 month from surgery
  In cases where microorganisms were identified in the wound culture results.
Wound bleeding | 1 month from surgery
  In cases where bleeding was visually observed from the wound or a hematoma was observed on the CT scan.
Wound dehiscence | 1 month from surgery
  In cases where the fascial closure was incomplete, causing part of the abdominal organs to protrude outside the abdomen, requiring surgical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

REFERENCES:
- [Derived] Pyo DH, Yun SH, Lee WY. A prospective single-arm clinical trial to assess the safety and efficacy of monofilament polydioxanone barbed suture, MONOFIX(R), on abdominal fascial closure. World J Surg. 2024 Jul;48(7):1674-1680. doi: 10.1002/wjs.12247. Epub 2024 Jun 15. PMID 38877993